CLINICAL TRIAL: NCT02719002
Title: Studying the Performance of OCT C-scan in the Screening for Retinopathy Related to Synthetic Antimalarials
Acronym: PERFOCTAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MMT_2015_45
Record Dates: First submitted 2016-03-16; First posted 2016-03-24 (Estimated); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Toxicity, Drug; Maculopathy
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Macular Degeneration

ARMS (1):
- OCT C-scan (Experimental)
  Interventions: Device: spectral domain optical coherence tomography C-scan and multifocal electroretinogram

INTERVENTIONS:
Device: spectral domain optical coherence tomography C-scan and multifocal electroretinogram

SUMMARY:
Maculopathy induced by retinal toxicity of synthetic antimalarials is to be screened at the sub-clinical stage. Indeed, when the first visual symptoms appear, macular damage is already irreversible and the clinical picture may even continue to deteriorate for several years after the end of synthetic antimalarial use. In opposition, the early termination of hydroxychloroquine in patients showing recent alterations on the multifocal electroretinogram (nfERG) allowed he reversibility of toxic damage over a six month period. It is therefore critical to detect early retinal anatomic changes during retinotoxicity screening before the occurrence of irreversible anatomical and functional consequences.

The usual patient monitoring consists of an annual eye examination, detecting subjective functional abnormalities (visual acuity, color vision, central visual field testing) or macular lesions (eye fundus). These abnormalities show a constituted infringement and do not contribute to the early diagnosis of synthetic antimalarial maculopathy.

The mfERG is an objective examination, able to detect retinal damage whilst still reversible. It is recommended during the annual monitoring and is, today, the gold standard for the screening and diagnosis of synthetic antimalarial maculopathy. However, its realization is time consuming, requires a good patient cooperation and is difficult to access due to the few ophthalmology centers offering it. In practice, it is rarely done as a systematic annual screening for patients on long-term synthetic antimalarial treatment. It is often limited to second-line studies (for patients already showing functional or anatomical abnormalities) whereas its interest lies in the detection of early lesions.

The Optical Coherence Tomography Spectral Domain (OCT-SD) is a non-invasive eye examination, commonly used since nearly 10 years. A special image analysis provides a panoramic viewing of the state of the photoreceptor layer, and a non-invasive detection of any anatomical changes, even subtle, within this layer.

The concordance between the "en face" OCT and the mfERG in the screening of synthetic antimalarial maculopathy is considered in this study.

ELIGIBILITY:
Inclusion Criteria:

* patients treated with synthetic antimalarials for at least 5 years

Exclusion Criteria:

* state of ocular structures preventing the realization of exams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
concordance between mfERG and SD OCT C-scan | 2 years
  measure of kappa coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmique Adolphe de Rothschild, Paris, France

REFERENCES:
- [Derived] Marques Dias JI, Chevalier K, Vasseur V, Laumonier E, Derrien S, Morel N, Le Guern V, Mathian A, Mouthon L, Mauget Faysse M, Nguyen Y, Costedoat-Chalumeau N. Comparison of flares in 85 patients with SLE who maintained, discontinued or reduced dose of hydroxychloroquine during a prospective study of ophthalmological screening for retinopathy (PERFOCTAPS Study). Lupus Sci Med. 2025 Mar 12;12(1):e001434. doi: 10.1136/lupus-2024-001434. PMID 40081891